

#### **Clinical Development**

PDR001, dabrafenib, trametinib

CPDR001F2301 / NCT02967692

A randomized, double-blind, placebo-controlled phase III study comparing the combination of PDR001, dabrafenib and trametinib versus placebo, dabrafenib and trametinib in previously untreated patients with unresectable or metastatic *BRAF* V600 mutant melanoma

# Statistical Analysis Plan (SAP) – Final and 5 year OS analysis

Document type: SAP Documentation

Document status: Final

Release date: 21-Aug-24

Number of pages: 16

Property of Novartis

Confidential

May not be used, divulged, published or otherwise disclosed without the consent of Novartis

# **Document History – Changes compared to previous final version of SAP**

| Date | Time<br>point | Reason<br>for<br>update | Outcome for update | Section and title impacted (Current) | ı |
|---|---|---|---|---|---|
| 21<br>August<br>2024 | Prior to<br>DB<br>lock | Creation<br>of final<br>version | To incorporate required analysis for OS and Safety. First Version. | relevant<br>required<br>analysis<br>final analy | een |

#### **Table of contents** 1 2 3 3.1 Efficacy......4 3.2 Exposure and Safety ......4 4 General Guidance for programming......5 5 References 16 6

#### 1 Introduction

This statistical analysis plan (SAP) describes all planned analyses for the five year follow-up overall survival (OS) and safety of **Part 1** (safety run-in), **Part 2** (Biomarker cohort) and **part 3** (randomized part) of the clinical study report (CSR) of study CPDR001F2301, a randomized, double-blind, placebo-controlled, phase III study comparing the combination of PDR001, dabrafenib and trametinib versus placebo, dabrafenib and trametinib in previously untreated patients with unresectable or metastatic *BRAF* V600 mutant melanoma. This will be also the final analysis for this study.

The content of this SAP is based on protocol CPDR001F2301 version 07 (Amendment 7, release date 27 Jan 2023). All decisions regarding follow-up analysis, as defined in the SAP document, have been made prior to database lock of the study data.

#### 2 Cut-off date

All analyses specified in this document will be conducted using the data from CPDR001F2301 study (cut-off date: 24Aug2024)

### 3 Statistical Analysis

Unless otherwise stated, all definitions and analysis methods are the same as given in the SAP used for the primary analysis of the study. Please refer to the final PFS analysis SAP for Part 3 (CPDR001F2301 Statistical Analysis Plan (SAP) for Part 3\_Amendment3\_Final) stored in CREDI dated 30-July-2020. And Part 1 and 2 ((CPDR001F2301 Statistical Analysis Plan (SAP) for Part 1 and 2\_Amendment3\_Final) stored in CREDI dated 30-July-2020.

The subject disposition will be summarized along with the overall survival and key safety endpoints for both Part 1 and 2 and Part 3 of the study separately.

Note: Any data entered after subject discontinued study due to any reason will be documented. However it will not be considered for analysis.

## 3.1 Efficacy

The following efficacy endpoints will be analyzed –

• Overall survival (OS)

All analyses will use the FAS, with no supportive analyses performed.

#### 3.2 Exposure and Safety

The following aspects will be summarized –

- Duration of exposure, dosing information and dose modifications will be summarized
- Overview of adverse events (number and % of subjects who died, with any AE, any SAE, any dose reductions/interruptions etc.), AEs by SOC and PT, summarized by relationship to study treatment (all AEs and AEs related to study treatment), seriousness

(SAEs and non-SAEs), AEs leading to treatment discontinuation and adverse events of special interest (AESI)

- Notable Vital Signs and ECG
- Deaths
- Hematology and Biochemistry laboratory data

## 4 General Guidance for programming

The same specification as in the TFL shells for Final PFS Analysis should be followed, unless otherwise specified as programming notes.

Note – The output numbers will be the same as to the primary CSR reporting activity.

## 5 List of outputs to be developed for this reporting activity

| Table number in final PFS CSR deliverables | Output title |
|---|---|
| Table 14.1-1.3 | Subject disposition (Full Analysis Set - Part 3) |
| Table 14.1-1.3b | Subject disposition (Full Analysis Set - Part 1 and 2) |
| Table 14.1-1.4 | Protocol deviations (Full Analysis Set - Part 3) |
| Table 14.1-1.4b | Protocol deviations (Full Analysis Set - Part 1 and 2) |
| Table 14.1-1.4a | Protocol deviations (Full Analysis Set - Part 3) – COVID-19 related PD's |
| Table 14.1-1.4a1 | Protocol deviations with relationship to COVID-19 (Full Analysis Set – Part 3) – COVID -19 related PD's |
| Table 14.1-3.8 | Post-treatment antineoplastic therapies by ATC class and preferred term (Full Analysis Set - Part 3) |
| Table 14.1-3.8b | Post-treatment antineoplastic therapies by ATC class and preferred term (Full Analysis Set - Part 1 and 2) |
| Table 14.1-3.9 | Post-treatment antineoplastic therapies by category (Full Analysis Set - Part 3) |
| Table 14.1-3.9b | Post-treatment antineoplastic therapies by category (Full Analysis Set - Part 1 and 2) |
| Table 14.1-3.10 | Summary of Best Overall Response on Subsequent Anti-<br>cancer therapy (Full Analysis Set – Part 3) |
| Figure 14.2-2.1 | Kaplan-Meier plot of Overall survival (OS) (months) (Full Analysis Set - Part 3) |
| Figure 14.2-2.1b | Kaplan-Meier plot of Overall survival (OS) (months) (Full Analysis Set - Part 1 and 2) |
| Figure 14.2-2.2 | Kaplan-Meier plot of Overall Survival (OS) (months) by stratification factors (Full Analysis Set - Part 3) |

| Figure 14.2-2.3 | Kaplan-Meier plot of Overall Survival (OS) (months) based on local investigator review and using RECIST 1.1 criteria – biomarker subgroups (Full Analysis Set - Part 3) |
|---|---|
| Figure 14.2-2.4 | Kaplan-Meier plot of Overall Survival (OS)(months) –Key subgroups of interest variables(Full Analysis Set - Part 3) |
| Figure 14.2-2.7 | Forest plot of Overall Survival (OS) (months) - Key subgroups of interest (Full Analysis Set - Part 3) |
| Figure 14.2-2.8 | Forest plot of Overall Survival (OS) (months) - Biomarker subgroups (Full Analysis Set - Part 3) |
| Figure 14.2-2.9 | Forest plot of Overall Survival (OS) (months) - Exploratory subgroups (Full Analysis Set - Part 3) |
| Table 14.2-2.6 | Stratified Piecewise Cox Regression analysis of Overall<br>Survival (OS) (months) (Full Analysis Set - Part 3) |
| Table 14.2-3.1 | Kaplan-Meier estimates of Overall Survival (OS) (months) (Full Analysis Set - Part 3) |
| Table 14.2-3.1a | Estimates of Overall Survival (OS) (months) (Full Analysis<br>Set - Part 3) – Sensitivity analysis based on COVID-19 |
| Table 14.2-3.1.1 | Kaplan-Meier estimates of Overall Survival (OS) (months)<br>(Pre-Protocol Set - Part 3) |
| Table 14.2-3.1b | Kaplan-Meier estimates of Overall Survival (OS) (months) (Full Analysis Set - Part 1 and 2) |
| Table 14.2-3.2 | Kaplan-Meier estimates of Overall Survival (OS) (months) by stratification factors (Full Analysis Set - Part 3) |
| Table 14.2-3.10 | Censoring reasons for Overall Survival (OS) (months) (Full Analysis Set - Part 3) |
| Table 14.2-3.10b | Censoring reasons for Overall Survival (OS) (months) (Full Analysis Set - Part 1 and 2) |
| Table 14.2-3.11 | Duration of follow-up (Full Analysis Set - Part 3) |
| Table 14.2-3.11b | Duration of follow-up (Full Analysis Set - Part 1 and 2) |
| Table 14.2-3.12 | Time on study (Full Analysis Set - Part 3) |
| Table 14.2-3.12b | Time on study (Full Analysis Set - Part 1 and 2) |
| Table 14.2-4.4 | Overall Survival (OS) (months) - Key subgroups (Full Analysis Set - Part 3) |
| Table 14.2-4.5 | Overall Survival (OS) (months) - Exploratory subgroups (Full Analysis Set - Part 3) |
| Table 14.2-4.6 | Overall Survival (OS) (months) - Biomarker subgroups (Full Analysis Set - Part 3) |
| Table 14.2-4.7 | Kaplan-Meier estimates of Overall Survival (OS) (months) by PD-L1 expression status (Full Analysis Set - Part 3) |
| Table 14.2-4.8 | Kaplan-Meier estimates of Overall Survival (OS)(months) by Cold tumors with lack of immunogenicity as defined by low TMB (< 10 mut/Mb) and low T-cell inflamed signature levels vs. all others (Full Analysis Set - Part 3) |

| Table 14.2-4.13 Kaplan-Meier estimates of Overall Survival (OS) (months) by TMB (Full Analysis Set - Part 3) Kaplan-Meier estimates of Overall Survival (OS) (months) by T-cell inflamed subgroups (Full Analysis Set - Part 3) Listing 14.2-2.6 Overall Survival (OS) (months) (Full Analysis Set - Part 3) eDISH plot: Peak total bilirubin vs Peak ALT and Peak AST (Safety set - Part 3) Table 14.3-1.1 Duration of exposure to PDR001/Placebo and summary of infusions (Safety Analysis Set - Part 3) Table 14.3-1.1b Duration of exposure to PDR001 and summary of infusions (Safety Analysis Set - Part 1 and 2) Duration of exposure to trametinib (Safety Analysis Set - Part 3) Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
|---|
| T-cell inflamed subgroups (Full Analysis Set - Part 3) Listing 14.2-2.6 Overall Survival (OS) (months) (Full Analysis Set - Part 3) Figure 14.3-1.6 eDISH plot: Peak total bilirubin vs Peak ALT and Peak AST (Safety set – Part 3) Table 14.3-1.1 Duration of exposure to PDR001/Placebo and summary of infusions (Safety Analysis Set - Part 3) Table 14.3-1.1b Duration of exposure to PDR001 and summary of infusions (Safety Analysis Set - Part 1 and 2) Table 14.3-1.2 Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
| Figure 14.3-1.6 eDISH plot: Peak total bilirubin vs Peak ALT and Peak AST (Safety set – Part 3) Duration of exposure to PDR001/Placebo and summary of infusions (Safety Analysis Set - Part 3) Table 14.3-1.1b Duration of exposure to PDR001 and summary of infusions (Safety Analysis Set - Part 1 and 2) Table 14.3-1.2 Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
| Table 14.3-1.0 Table 14.3-1.1 Table 14.3-1.1b Table 14.3-1.1b Table 14.3-1.1b Table 14.3-1.2 Table 14.3-1.2 Ouration of exposure to PDR001/Placebo and summary of infusions (Safety Analysis Set - Part 3) Duration of exposure to PDR001 and summary of infusions (Safety Analysis Set - Part 1 and 2) Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
| Table 14.3-1.1 infusions (Safety Analysis Set - Part 3) Table 14.3-1.1b Duration of exposure to PDR001 and summary of infusions (Safety Analysis Set - Part 1 and 2) Table 14.3-1.2 Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
| (Safety Analysis Set - Part 1 and 2) Table 14.3-1.2 Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
| Table 14.3-1.2 Duration of exposure to trametinib (Safety Analysis Set - Part 3) |
| T 11 14 2 1 21 D 2 C 2 |
| Table 14.3-1.2b Duration of exposure to trametinib (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-1.3 Duration of exposure to dabrafenib (Safety Analysis Set - Part 3) |
| Table 14.3-1.3b Duration of exposure to dabrafenib (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-1.4 Duration of exposure to study treatment (Safety Analysis Set - Part 3) |
| Table 14.3-1.4b Duration of exposure to study treatment (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-2.1 Dose of PDR001/Placebo received (Safety Analysis Set - Part 3) |
| Table 14.3-2.1b Dose of PDR001 received (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-2.2 Dose of trametinib received (Safety Analysis Set - Part 3) |
| Table 14.3-2.2b Dose of trametinib received (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-2.3 Dose of dabrafenib received (Safety Analysis Set - Part 3) |
| Table 14.3-2.3b Dose of dabrafenib received (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-2.5 Dose adjustments and discontinuation of PDR001/Placebo (Safety Analysis Set - Part 3) |
| Table 14.3-2.5b Dose adjustments and discontinuation of PDR001 (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-2.6 Dose adjustments and discontinuation of dabrafenib (Safety Analysis Set - Part 3) |
| Table 14.3-2.6b Dose adjustments and discontinuation of dabrafenib (Safety Analysis Set - Part 1 and 2) |

| Table 14.3-2.7 | Dose adjustments and discontinuation of trametinib (Safety Analysis Set - Part 3) |
|---|---|
| Table 14.3-2.7b | Dose adjustments and discontinuation of trametinib (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-3.4 | Concomitant medications by ATC class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3-3.4b | Concomitant medications by ATC class and preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-3.4.1 | Concomitant medications by ATC class and preferred term -<br>Extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3-3.4.1b | Concomitant medications by ATC class and preferred term -<br>Extended follow-up (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-3.7 | Concomitant medications with immunosuppressive intent by preferred term (Safety Analysis Set - Part 3) |
| Table 14.3-3.7b | Concomitant medications with immunosuppressive intent by preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-3.8 | Concomitant medications with immunosuppressive intent by preferred term - Extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3-3.8b | Concomitant medications with immunosuppressive intent by preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.1 | Worst post-baseline biochemistry abnormalities based on CTC grades (Safety Analysis Set - Part 3) |
| Table 14.3-5.1b | Worst post-baseline biochemistry abnormalities based on CTC grades (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.2 | Worst post-baseline hematology abnormalities based on CTC grades (Safety Analysis Set - Part 3) |
| Table 14.3-5.2b | Worst post-baseline hematology abnormalities based on CTC grades (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.4 | Hematology shift table based on CTC grades (Safety Analysis Set - Part 3) |
| Table 14.3-5.4b | Hematology shift table based on CTC grades (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.5 | Biochemistry shift table based on CTC grades (Safety Analysis Set - Part 3) |
| Table 14.3-5.5b | Biochemistry shift table based on CTC grades (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.6 | Hematology shift table based on normal ranges (Safety Analysis Set - Part 3) |
| Table 14.3-5.6b | Hematology shift table based on normal ranges (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.7 | Biochemistry shift table based on normal ranges (Safety<br>Analysis Set - Part 3) |

| Table 14.3-5.7b | Biochemistry shift table based on normal ranges (Safety Analysis Set - Part 1 and 2) |
|---|---|
| Table 14.3-5.8 | Summary of hepatic laboratory values (Safety Analysis Set - Part 3) |
| Table 14.3-5.8b | Summary of hepatic laboratory values (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.10 | Notable ECG values (Safety Analysis Set - Part 3) |
| Table 14.3-5.10b | Notable ECG values (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.11 | Shift tables of ECOG performance status from baseline to worst post-baseline ECOG status by score (Safety Analysis Set - Part 3) |
| Table 14.3-5.11b | Shift tables of ECOG performance status from baseline to worst post-baseline ECOG status by score (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.12 | Shift tables of ECOG performance status from baseline to best post-baseline ECOG status by score (Safety Analysis Set - Part 3) |
| Table 14.3-5.12b | Shift tables of ECOG performance status from baseline to best post-baseline ECOG status by score (Safety Analysis Set - Part 1 and 2) |
| Table 14.3-5.15 | Notable vital sign values (Safety Analysis Set - Part 3) |
| Table 14.3-5.15b | Notable vital sign values (Safety Analysis Set – Part 1 and 2) |
| Table 14.3-5.16 | Change from baseline vital signs by timepoint (Safety Analysis Set - Part 3) |
| Table 14.3-5.16b | Change from baseline vital signs by timepoint (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.1.2 | Overview of adverse events (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.1.2b | Overview of adverse events (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.1.3 | Overview of adverse events - Extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.1.3b | Overview of adverse events - Extended follow-up (Safety Analysis Set - Part 1 and 2 |
| Table 14.3.1-1.2.2 | Adverse events by preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.2.2b | Adverse events by preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.2.2a | Adverse events by preferred term (Safety Analysis Set - Part 3) - Non-specific COVID -19 related terms(pre-COVID period) |
| Table 14.3.1-1.2.2a1 | Adverse events by preferred term (Safety Analysis Set - Part 3) – Non-specific COVID -19 related terms(Complete study period) |
| Table 14.3.1-<br>1.2.2a2 | Adverse events by preferred term (Safety Analysis Set - Part 3) – specific COVID -19 related terms |

| Table 14.3.1-1.2.3 | Adverse events by system organ class and preferred term |
|---|---|
| | (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.2.3b | Adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) |
| T 11 1421124 | Adverse events by system organ class and preferred term - |
| Table 14.3.1-1.2.4 | extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.2.4b | Adverse events by system organ class and preferred term - |
| | extended follow-up (Safety Analysis Set - Part 1 and 2) |
| | Adverse events suspected to be study treatment related by |
| Table 14.3.1-1.2.7 | system organ class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.2.7b | Adverse events suspected to be study treatment related by |
| | system organ class and preferred term (Safety Analysis Set - |
| | Part 1 and 2) |
| | Adverse events suspected to be study treatment related by |
| Table 14.3.1-1.2.8 | system organ class and preferred term - Extended follow-up |
| T 11 14 2 1 1 2 01 | (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.2.8b | Adverse events suspected to be study treatment related by |
| | system organ class and preferred term - Extended follow-up |
| | (Safety Analysis Set - Part 1 and 2) Treatment-related adverse events by preferred term (Safety |
| Table 14.3.1-1.2.9 | Analysis Set - Part 3) |
| T-1.1. 14211201 | |
| Table 14.3.1-1.2.9b | Treatment-related adverse events by preferred term (Safety |
| 1able 14.3.1-1.2.90 | Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.2.96 Table 14.3.1-1.3.1 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) |
| | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set |
| Table 14.3.1-1.3.1 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.1b | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.1b | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.1b Table 14.3.1-1.3.2 Table 14.3.1-1.3.2b | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.1b Table 14.3.1-1.3.2 Table 14.3.1-1.3.2b | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 Table 14.3.1-1.3.3 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 Table 14.3.1-1.3.3 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome (Safety Analysis Set |
| Table 14.3.1-1.3.1 Table 14.3.1-1.3.1b Table 14.3.1-1.3.2 Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 Table 14.3.1-1.3.3b Table 14.3.1-1.3.4 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome (Safety Analysis Set - Part 3) Serious adverse events with fatal outcome (Safety Analysis Set - Part 3) Serious adverse events with fatal outcome (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 Table 14.3.1-1.3.3b Table 14.3.1-1.3.4b Table 14.3.1-1.3.4 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome (Safety Analysis Set - Part 3) Serious adverse events with fatal outcome (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome - Extended Follow-serious adve |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 Table 14.3.1-1.3.3b Table 14.3.1-1.3.4b Table 14.3.1-1.3.4b Table 14.3.1-1.3.5 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome (Safety Analysis Set - Part 3) Serious adverse events with fatal outcome (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome - Extended Follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.3.1b Table 14.3.1-1.3.2b Table 14.3.1-1.3.2b Table 14.3.1-1.3.3 Table 14.3.1-1.3.3b Table 14.3.1-1.3.4b Table 14.3.1-1.3.4 | Analysis Set - Part 1 and 2) Serious adverse events by preferred term (Safety Analysis Set - Part 3) Serious adverse events by preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 3) Serious adverse events by system organ class and preferred term - Extended follow-up (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome (Safety Analysis Set - Part 3) Serious adverse events with fatal outcome (Safety Analysis Set - Part 1 and 2) Serious adverse events with fatal outcome - Extended Follow-serious adve |

| Table 14.3.1-1.3.6 | Serious adverse events with fatal outcome - Key subgroups |
|---|---|
| Table 14.3.1-1.3.7 | (Safety Analysis Set - Part 3) Serious adverse events with fatal outcome - Extended Follow- |
| | up - Key subgroups (Safety Analysis Set - Part 3) Serious adverse events suspected to be study treatment related |
| Table 14.3.1-1.3.8 | by system organ class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.3.9 | Serious adverse events suspected to be study treatment related<br>by system organ class and preferred term - Extended follow-up<br>(Safety Analysis Set - Part 3) |
| Table 14.3.1-1.3.9b | Serious adverse events suspected to be study treatment related<br>by system organ class and preferred term - Extended follow-up<br>(Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.4.1 | Adverse events leading to treatment discontinuation by preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.4.1b | Adverse events leading to treatment discontinuation by preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.4.2 | Adverse events leading to study treatment discontinuation, regardless of study treatment relationship by system organ class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.4.2b | Adverse events leading to study treatment discontinuation, regardless of study treatment relationship by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.4.3 | Adverse events leading to study treatment discontinuation, suspected to be study treatment related by system organ class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1-1.4.3b | Adverse events leading to study treatment discontinuation, suspected to be study treatment related by system organ class and preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.12.1 | All Deaths (Safety Analysis Set - Part 3) |
| Table 14.3.1-<br>1.12.1b | All Deaths (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.13.1 | Non-serious adverse events (threshold = 5%) by system organ class and preferred term (Safety Analysis Set - Part 3) |
| Table 14.3.1- | Non-serious adverse events (threshold = 5%) by system organ |
| 1.13.1b | class and preferred term (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-1.13.2 | Non-serious adverse events (threshold = 5%) by system organ class and preferred term including extended safety follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-<br>1.13.2b | Non-serious adverse events (threshold = 5%) by system organ class and preferred term including extended safety follow-up (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.1.1 | Overview of adverse events of special interest for PDR001 (Safety Analysis Set - Part 3) |

| Table 14.3.1-2.1.1b | Overview of adverse events of special interest for PDR001 (Safety Analysis Set - Part 1 and 2) |
|---|---|
| Table 14.3.1-2.1.2 | Overview of adverse events of special interest for PDR001 -<br>Extended follow-up (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.1.2b | Overview of adverse events of special interest for PDR001 - Extended follow-up (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.3.1 | Overview of serious adverse events of special interest for PDR001 (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.3.1b | Overview of serious adverse events of special interest for PDR001 (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.3.3 | Overview of serious adverse events of special interest for dabrafenib and trametinib (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.3.3b | Overview of serious adverse events of special interest for dabrafenib and trametinib (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.5.1 | Overview of adverse events of special interest for combination of dabrafenib and trametinib (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.5.1b | Overview of adverse events of special interest for combination of dabrafenib and trametinib (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.6.1 | Overview of adverse events of special interest for PDR001 leading to treatment discontinuation (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.6.1b | Overview of adverse events of special interest for PDR001 leading to treatment discontinuation (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.7.1 | Overview of adverse events of special interest for PDR001 requiring immunosuppressive medication (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.8.1b | Overview of adverse events of special interest for PDR001 requiring immunosuppressive medication (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.9.1 | Overview of adverse events of special interest for PDR001 leading to dose adjustment/interruption (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.9.1b | Overview of adverse events of special interest for PDR001 leading to dose adjustment/interruption (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.10.1 | Overview of adverse events of special interest for dabrafenib<br>and trametinib leading to dose adjustment/interruption of<br>dabrafenib or trametinib (Safety Analysis Set - Part 3) |
| Table 14.3.1-2.10.1b | Overview of adverse events of special interest for dabrafenib and trametinib leading to dose adjustment/interruption of dabrafenib or trametinib (Safety Analysis Set - Part 1 and 2) |
| Table 14.3.1-2.11.1 | Overview of adverse events of special interest for PDR001 leading to death (Safety Analysis Set - Part 3) |

| 001 |
|------------------|
| fenib<br>art 3) |
| fenib |
| art 1 |
| 001 |
| lnisone |
| 001 |
| lnisone |
| 001 |
| lnisone |
| 001 |
| lnisone |
| ination |
| steroid |
| lysis |
| • .• |
| ination |
| steroid |
| lysis |
| · |
| ination |
| steroid |
| lysis |
| ination |
| rtaroid |
| steroid |
| steroid<br>lysis |
| lysis<br>Part 3) |
| lysis |
| Part 3) |
| lysis<br>Part 3) |
| Part 3) |
| Part 3) Part 1 |
| Part 3) Part 1 |

| Table 14.3.1-2.15.6 | Grade 3 or higher AESIs by month of occurrence (Safety Analysis Set - Part 3 |
|---|---|
| Table 14.3.1-3.1.1 | Summary of event of pyrexia (Preferred Term) (Safety Analysis Set - Part 3) |
| Table 14.3.1-3.1.1b | Summary of event of pyrexia (Preferred Term) (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-1.1 | Deaths (Safety Analysis Set - Part 3) |
| Listing 14.3.2-1.1a | Deaths – COVID-19 related (Safety Analysis Set - Part 3) |
| Listing 14.3.2-1.1b | Deaths (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-<br>1.1b1 | Deaths – COVID-19 related (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-1.4 | Adverse events leading to discontinuation (Safety Analysis Set - Part 3) |
| Listing 14.3.2-1.4b | Adverse events leading to discontinuation (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-1.5 | Adverse events leading to dose adjustment and/or interruption (Safety Analysis Set - Part 3) |
| Listing 14.3.2-1.5b | Adverse events leading to dose adjustment and/or interruption (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-1.6 | Serious adverse events (Safety Analysis Set - Part 3) |
| Listing 14.3.2-1.6b | Serious adverse events (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-1.7 | Serious adverse events with fatal outcome (Safety Analysis Set - Part 3) |
| Listing 14.3.2-1.7b | Serious adverse events with fatal outcome (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-2.1 | Adverse events of special interest of PDR001 (Safety Analysis Set - Part 3) |
| Listing 14.3.2-2.1b | Adverse events of special interest of PDR001 (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.2-2.2 | Adverse events of special interest for combination of dabrafenib and trametinib (Safety Analysis Set - Part 3) |
| Listing 14.3.2-2.2b | Adverse events of special interest for combination of dabrafenib and trametinib (Safety Analysis Set - Part 1 and 2) |
| Listing 14.3.4-1.1 | Subjects with notable ECG values (Safety Analysis Set - Part 3) |
| Listing 14.3.4-1.1b | Subject with notable ECG values (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.1-1.1 | Subject disposition (Full Analysis Set - Part 3) |
| Listing 16.2.1-1.1b | Subject disposition (Full Analysis Set - Part 1 and 2) |
| Listing 16.2.2-1.1 | Protocol deviations (Full Analysis Set - Part 3) |
| Listing 16.2.2-1.1b | Protocol deviations (Full Analysis Set - Part 1 and 2) |
| Listing 16.2.2-1.1a | Protocol deviations (Full Analysis Set - Part 3) – COVID-19 related PD's |

| Listing 16.2.2-<br>1.1b1 | Protocol deviations (Full Analysis Set - Part 1 and 2) – COVID-19 related PD's |
|---|---|
| Listing 16.2.4-5.5 | Post treatment antineoplastic therapy – Surgery (Full Analysis Set - Part 3) |
| Listing 16.2.4-5.5b | Post treatment antineoplastic therapy – Surgery (Full Analysis Set - Part 1 and 2) |
| Listing 16.2.4-5.6 | Post treatment antineoplastic therapy – Radiotherapy (Full Analysis Set - Part 3) |
| Listing 16.2.4-5.6b | Post treatment antineoplastic therapy – Radiotherapy (Full Analysis Set - Part 1 and 2) |
| Listing 16.2.4-5.7 | Post treatment antineoplastic therapy – Medications (Full Analysis Set - Part 3) |
| Listing 16.2.4-5.7b | Post treatment antineoplastic therapy – Medications (Full Analysis Set - Part 1 and 2) |
| Listing 16.2.5-1.1 | Dose administration record for PDR001/Placebo (Safety Analysis Set - Part 3) |
| Listing 16.2.5-1.1b | Dose administration record for PDR001 (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.5-1.2 | Dose administration record for Dabrafenib (Safety Analysis Set - Part 3) |
| Listing 16.2.5-1.2b | Dose administration record for dabrafenib (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.5-1.3 | Dose administration record for Trametinib (Safety Analysis Set - Part 3) |
| Listing 16.2.5-1.3b | Dose administration record for trametinib (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.7-1.2 | Adverse events (Safety Analysis Set - Part 3) |
| Listing 16.2.7-1.2b | Adverse events (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.7- | Adverse events (Safety Analysis Set - Part 1 and 2) – COVID- |
| 1.2b1 | 19 related |
| Listing 16.2.7-1.2a | Adverse events (Safety Analysis Set - Part 3) – Specific COVID-19 related |
| Listing 16.2.7- | Adverse events (Safety Analysis Set - Part 3) – Non-Specific |
| 1.2a1 | COVID-19 related (Complete study period) |
| Listing 16.2.7-2.2 | Infusion Reaction Related Adverse Events of AESI after Dose (Safety Analysis Set - Part 3) |
| Listing 16.2.7-2.2b | Infusion Reaction Related Adverse Events of AESI after Dose (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.8-1.1 | Subject with CTC grade 3 or 4 laboratory values (Safety Analysis Set - Part 3) |
| Listing 16.2.8-1.1b | Subject with CTC grade 3 or 4 laboratory values (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.8-1.2 | Subject laboratory profile: Hematology (Safety Analysis Set - Part 3) |

| Listing 16.2.8-1.2b | Subject laboratory profile: Hematology (Safety Analysis Set - Part 1 and 2) |
|---|---|
| Listing 16.2.8-1.3 | Subject laboratory profile: Biochemistry (Safety Analysis Set - Part 3) |
| Listing 16.2.8-1.3b | Subject laboratory profile: Biochemistry (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.8-1.4 | Subject laboratory profile of hepatic laboratory values (Safety Analysis Set - Part 3) |
| Listing 16.2.8-1.4b | Subject laboratory profile of hepatic laboratory values (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.9-1.1 | Subjects with notable Vital signs (Safety Analysis Set - Part 3) |
| Listing 16.2.9-1.1b | Subjects with notable Vital signs (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.9-2.1 | ECOG performance status (Safety Analysis Set - Part 3) |
| Listing 16.2.9-2.1b | ECOG performance status (Safety Analysis Set - Part 1 and 2) |
| Listing 16.2.9-4.1 | Cardiac imaging (Safety Analysis Set - Part 3) |
| Listing 16.2.9-4.1b | Cardiac imaging (Safety Analysis Set - Part 1 and 2) |

## 6 References

- 1. Protocol amendment 7, release date 27 Jan 2023
- 2. SAP used for the primary analysis of the study.







CPDR001F2301 TFL CPDR001F2301 CPDR001F2301 for final PFS analysisStatistical Analysis PStatistical Analysis P